CLINICAL TRIAL: NCT05743192
Title: Discontinuation of Antibiotic Susceptibility Testing on Monobacterial Enterococcus Faecalis Positive Urine Cultures: an Impact on Antibiotic Prescriptions?
Brief Title: Discontinuation of Antibiotic Susceptibility Testing on Enterococcus Faecalis Positive Urine Cultures in Hospitalized Patients: an Impact on Antibiotic Prescriptions? (FaecaCible)
Acronym: FaecaCible
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BARONNET Guillaume, MD, Infectious diseases department, Central Hospital, Nancy, France
Other Study IDs: 2022PI075
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Antibiotic Susceptibility Reporting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before group: Group of patients with a positive urine culture for Enterococcus faecalis before the procedure consisting of systematically performing an antibiotic susceptibility test.
- After group: Group of patients with a positive urine culture for Enterococcus faecalis after the procedure consisting of systematically performing an antibiotic susceptibility test.
  Interventions: Other: Stop performing an antibiotic susceptibility test

INTERVENTIONS:
Other: Stop performing an antibiotic susceptibility test — Intervention = Stop performing an antibiotic susceptibility test for enterococcus faecalis in urine cultures. It defines two groups : one before and one after the intervention
  Groups: After group

SUMMARY:
The objective of the study is to evaluate the impact of not reporting antibiotic susceptibility tests on antibiotic consumption for Enterococcus faecalis positive urine cultures in adult hospitalized patients. The secondary objectives are to evaluate the impact of this intervention on antibiotic prescription rates as well as on antibiotic consumption according to: patient gender, type of antibiotic therapy (probabilistic/documented) and diagnosis (urinary tract infection or colonization). It is hypothesized that antibiotic consumption is lower after the application of the absence of antibiotic susceptibility reporting compared to before.

ELIGIBILITY:
Inclusion Criteria:

* Person having received complete information on the organization of the research and not having objected to the exploitation of these data
* Adult patients (More than 18);
* Having performed a urine culture at the Nancy University Hospital, taken from the 2nd urine stream, by urinary catheter or via a suprapubic catheter and whose culture is positive for monomicrobial E. faecalis with a bacteriuria threshold greater than or equal to 10^3 CFU/field;
* Hospitalized at the Nancy University Hospital at least 72 hours after validation of the antibiotic susceptibility test in the pre-intervention period and at least 72 hours after validation of the culture in the post-intervention period.

Exclusion Criteria:

* Inpatients in hematology, critical care/intensive care, consultation and day hospital units;
* Urine cultures performed in ambulatory units ;
* Urine culture performed in the critical care/intensive care/hematology units;
* Patients discharged from hospital/deceased/transferred to intensive care within 72 hours of the validation of the antibiotic susceptibility test or the validation of the urine culture;
* Patients with associated E. faecalis bacteremia;
* Urine culture without an antibiotic susceptibility test for the pre-intervention period;
* Urine culture with a monomicrobial history of less than 1 week;
* Culture of urine from pyelic punctures or nephrostomy tubes - conservation of those from second streams, urinary catheters and suprapubic catheters).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These are urine cultures taken from 2nd urine stream, by urinary catheter or via a suprapubic catheter and with a positive culture for monomicrobial Enterococcus faecalis with a bacteriuria threshold greater than or equal to 10^3. These urine cultures were performed between December 10, 2018 and December 10, 2020 in adults hospitalized at the Nancy University Hospital and present at least 72 hours after the validation of the antibiogram or the identification of the germ, excluding hospitalization or passage in hematology services, continuous care/intensive care, day hospitalization and consultation.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Proportion of positive urine culture for which antibiotic therapy was prescribed (%) | Between 24 hours before the urine culture is collected and 72 hours following the validation of the antibiotic susceptibility test/the urine culture by the biologist

SECONDARY OUTCOMES:
Prescription rate of each antibiotic class/molecule (%) | Between 24 hours before the urine culture is collected and 72 hours following the validation of the antibiotic susceptibility test/the urine culture by the biologist
Proportion of urine cultures for which antibiotic therapy was prescribed (%) by type of antibiotic therapy. | Between 24 hours before the urine culture is collected and 72 hours following the validation of the antibiotic susceptibility test/the urine culture by the biologist
  Type of antibiotic therapy = probabilistic or documented
Prescription rate of each antibiotic class/molecule (%) by type of antibiotic therapy. | Between 24 hours before the urine culture is collected and 72 hours following the validation of the antibiotic susceptibility test/the urine culture by the biologist
Proportion of urine cultures for which antibiotic therapy was prescribed (%) by sex of patient | Between 24 hours before the urine culture is collected and 72 hours following the validation of the antibiotic susceptibility test/the urine culture by the biologist
Prescription rate of each antibiotic class/molecule (%) by patient gender | Between 24 hours before the urine culture is collected and 72 hours following the validation of the antibiotic susceptibility test/the urine culture by the biologist
Proportion of urine cultures for which antibiotic therapy was prescribed (%) by diagnosis | Between 24 hours before the urine culture is collected and 72 hours following the validation of the antibiotic susceptibility test/the urine culture by the biologist
  Diagnosis = UTI or UCC
Prescription rate of each antibiotic class/molecule (%) by diagnosis | Between 24 hours before the urine culture is collected and 72 hours following the validation of the antibiotic susceptibility test/the urine culture by the biologist
  Diagnosis = UTI or UCC

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy University Hospital, Vandœuvre-lès-Nancy, France